CLINICAL TRIAL: NCT01383356
Title: A Single Dose Comparative Bioavailability Study of Linagliptin/Metformin hydrochloride2.5mg/500mg Combination Tablets Versus Linagliptin 2.5mg Tablets Administered With Glucophage 500mg Tablets Under Fasting Conditions
Brief Title: Comparison of the Bioavailability of Metformin Between Medium Dose Linagliptin/Metformin Tablets and Medium Dose Glucophage Tablet Given With Linagliptin Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1288.19
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin/Metformin medium dosecombo (Experimental): patient to receive a single medium dose combination tablet containing Linagliptin and Metformin once daily
  Interventions: Drug: Linagliptin/Metformin Combo
- Linagliptin plus Metformin medium dose (Active Comparator): patient to receive two individual tablets: Linagliptin and Metformin (medium dose)
  Interventions: Drug: Metformin Single Tablet; Drug: Linagliptin Single Tablet

INTERVENTIONS:
Drug: Metformin Single Tablet — Metformin medium doseTablet
  Arms: Linagliptin plus Metformin medium dose
Drug: Linagliptin/Metformin Combo — Fixed dose combination
  Arms: Linagliptin/Metformin medium dosecombo
Drug: Linagliptin Single Tablet — Linagliptin Single medium dose Tablet
  Arms: Linagliptin plus Metformin medium dose

SUMMARY:
The data from this study will be used to compare the kinetic profile of metformin 500mg in linagliptin/metformin fixed dose combination tablet versus Canadian metformin reference product administered concomitantly with linagliptin 2.5 mg tablet.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects.

Exclusion criteria:

1. Any relevant deviation from healthy conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.19.1 Boehringer Ingelheim Investigational Site, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 subjects were enrolled in the original study (June 2011 to July 2011) and 40 in the add-on study (November 2011 to December 2011) which was an option provided by protocol to increase the subject number. As no significant STUDY and STUDY-by-TREATMENT effect was revealed in analysis of pooled data, final analysis was performed on pooled data.
Pre-assignment Details: This is a 2 period, 2 sequence, 2 treatment crossover. Subjects were randomized to one of the two sequences AB or BA. The duration of washout was at least 35 days between dosing.
Groups:
- Lina/Met 2.5mg/500mg Then Lina 2.5mg Plus Met 500mg: Combination tablet Linagliptin (Lina) /Metformin (Met) 2.5mg/500mg followed by single tablets Linagliptin 2.5mg plus Metformin 500mg
- Lina 2.5mg Plus Met 500mg Then Lina/Met 2.5mg/500mg: Single tablets Linagliptin 2.5mg plus Metformin 500mg followed by combination tablet Linagliptin/Metformin 2.5mg/500mg
Period: Period 1
Arm/Group | Lina/Met 2.5mg/500mg Then Lina 2.5mg Plus Met 500mg | Lina 2.5mg Plus Met 500mg Then Lina/Met 2.5mg/500mg
Started | 29 (Entered and treated.) | 29 (Entered and treated.)
Completed | 21 (Completed period 1.) | 23 (Completed period 1.)
Not Completed | 8 | 6
Not completed — Adverse Event | 5 | 3
Not completed — Non-compliance | 3 | 0
Not completed — Out of Range Mid-study-Test | 0 | 1
Not completed — Personal | 0 | 2
Period: Washout Period (at Least 35 Days)
Arm/Group | Lina/Met 2.5mg/500mg Then Lina 2.5mg Plus Met 500mg | Lina 2.5mg Plus Met 500mg Then Lina/Met 2.5mg/500mg
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Lina/Met 2.5mg/500mg Then Lina 2.5mg Plus Met 500mg | Lina 2.5mg Plus Met 500mg Then Lina/Met 2.5mg/500mg
Started | 21 (Entered and treated.) | 23 (Entered and treated.)
Completed | 21 (Completed period 2.) | 23 (Completed period 2.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dosed participants from combined studies
Groups:
- Entire Study Population: Total number of subjects randomised and treated in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum measured concentration of metformin in plasma, per period.
Time Frame: Prior to drug administration and at 0.33, 0.67, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 30, and 36 hours post dose in each treatment period
Population: All subjects having all samples in all periods and subjects who missed samples that may not affect the estimation of pharmacokinetic parameters in any period.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Lina/Met 2.5mg/500mg: Combination tablet
- Lina 2.5mg Plus Met 500mg: Single tablets
Arm/Group | Lina/Met 2.5mg/500mg | Lina 2.5mg Plus Met 500mg
Number analyzed (Participants) | 44 | 44
ng/ml | 901.82 (262.45) | 770.52 (189.44)
Statistical Analysis 1: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; The two formulations are shown to be bioequivalent if the geometric mean ratio is contained within the 80 to 125 percent range both on measured data (statistical analysis 1) and on potency corrected data (percent potency of label claim) (statistical analysis 2). ANOVA was applied to log-transformed Cmax and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction; Test type: Non-Inferiority or Equivalence — Bioequivalence; Geometric mean ratio (GMR) in percent = 118, 90% CI 2-sided [111 to 125] — Lina/Met 2.5mg/500mg versus (vs.) Lina 2.5mg plus Met 500mg
Statistical Analysis 2: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; ANOVA was applied to log-transformed Cmax and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction. Results were potency corrected (GMR multiplied by the quotient of drug potency (DP) of Met in single tablet and DP of Met in combination tablet); Test type: Non-Inferiority or Equivalence — Bioequivalence; GMR, potency corrected (percent) = 122, 90% CI 2-sided [114 to 130] — Lina/Met 2.5mg/500mg vs. Lina 2.5mg plus Met 500mg

2. Primary Outcome: Area Under the Curve 0 to Last Measurable Value (AUC0-t)
Description: AUC0-t is the area under the concentration versus time curve of metformin in plasma, from time zero (0) to the time of the last measurable analyte concentration (t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Lina/Met 2.5mg/500mg | Lina 2.5mg Plus Met 500mg
Number analyzed (Participants) | 44 | 44
ng*h/ml | 7079.65 (1688.14) | 6808.27 (1708.20)
Statistical Analysis 1: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; The two formulations are shown to be bioequivalent if the 90 percent confidence interval of geometric mean ratio is entirely contained within the 80 to125 percent range both on measured data (statistical analysis 1) and potency corrected data (percent potency of label claim) (statistical analysis 2). ANOVA was applied to log-transformed AUC0-t and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction; Test type: Non-Inferiority or Equivalence — Bioequivalence; Geometric mean ratio (percent) = 105, 90% CI [101 to 108] — Lina/Met 2.5mg/500mg vs. Lina 2.5mg plus Met 500mg
Statistical Analysis 2: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; ANOVA was applied to log-transformed AUC0-t and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction. Results were potency corrected (GMR multiplied by the quotient of DP of Met in single tablet and DP of Met in combination tablet); Test type: Non-Inferiority or Equivalence — Bioequivalence; GMR, potency corrected (percent) = 108, 90% CI [105 to 112] — Lina/Met 2.5mg/500mg vs.Lina 2.5mg plus Met 500mg

3. Secondary Outcome: Area Under the Curve 0 to Inf (AUC0-inf)
Description: AUC0-inf is the area under the concentration versus time curve of metformin in plasma from time zero extrapolated to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Lina/Met 2.5mg/500mg | Lina 2.5mg Plus Met 500mg
Number analyzed (Participants) | 44 | 44
ng*h/ml | 7198.79 (1689.89) | 6923.79 (1714.08)
Statistical Analysis 1: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; ANOVA was applied to log-transformed AUC0-inf and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction; Test type: Non-Inferiority or Equivalence — Bioequivalence (BE), AUC0-inf was no BE criteria; Geometric mean ratio (percent) = 105, 90% CI [101 to 108] — Lina/Met 2.5mg/500mg vs. Lina 2.5mg plus Met 500mg
Statistical Analysis 2: Comparison: Lina/Met 2.5mg/500mg vs Lina 2.5mg Plus Met 500mg; ANOVA was applied to log-transformed AUC0-inf and included study, subject-within-study, period-within-study, treatment and study-by-treatment interaction. Results were potency corrected (GMR multiplied by the quotient of DP of Met in single tablet and DP of Met in combination tablet); Test type: Non-Inferiority or Equivalence — BE, AUC0-inf was no BE criteria; GMR, potency corrected (percent) = 108, 90% CI [105 to 112] — Lina/Met 2.5mg/500mg vs. Lina 2.5mg plus Met 500mg

ADVERSE EVENTS:
Time Frame: Period 1 (36 hours)+ Washout (35 days) +Period 2 (36 hours)
Arm/Group | Lina/Met 2.5mg/500mg | Lina 2.5mg Plus Met 500mg
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 17/52 | 21/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lina/Met 2.5mg/500mg (N=52) | Lina 2.5mg Plus Met 500mg (N=50)
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 9 | 8
Vomiting (Gastrointestinal disorders) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Dizziness (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.